CLINICAL TRIAL: NCT06843317
Title: A Phase 1, Placebo-controlled, Randomized, Observer-blind Study to Describe the Safety, Tolerability and Immunogenicity of SCB-1019T in Adults Who Were Vaccinated With AREXVY at Least 18 Months Before
Brief Title: Safety and Immunogenicity Study of Revaccination With SCB-1019T in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals USA, LLC (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-1019-002
Record Dates: First submitted 2025-02-20; First posted 2025-02-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — arexvy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (SCB-1019T) (Experimental): 50 adults to receive low dose SCB-1019T at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019T
- Group 2 (SCB-1019T) (Experimental): 50 adults to receive high dose SCB-1019T at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019T
- Group 3 (AREXVY) (Active Comparator): 50 adults to receive AREXVY at Day 1
  Interventions: Biological: AREXVY
- Group 4 (Placebo) (Placebo Comparator): 10 adults to receive Placebo at Day 1
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Candidate vaccine, SCB-1019T — SCB-1019T is a novel bivalent recombinant RSV vaccine (CHO Cell) designed to broadly neutralize the two dominant circulating strains of the virus. The SCB-1019T vaccine consists of the PreF protein subunits from the two dominant circulating strains, strain A and strain B, fused to Trimer-Tag™.
  Arms: Group 1 (SCB-1019T); Group 2 (SCB-1019T)
Biological: AREXVY — positive comparator
  Arms: Group 3 (AREXVY)
Other: placebo — Placebo Comparator
  Arms: Group 4 (Placebo)

SUMMARY:
CLO-SCB-1019-002 is the first study of SCB-1019T vaccine for revaccination in older adults who were previously vaccinated with AREXVY. The safety, tolerability and immunogenicity of SCB-1019T are assessed.

DETAILED DESCRIPTION:
The study design will compare heterologous revaccination with SCB-1019T, homologous revaccination with AREXVY, or placebo in adults who were previously vaccinated with AREXVY. The sample size for this study is not based on formal statistical hypothesis testing but is acceptable for safety and immunogenicity evaluation in a phase 1 study. The study will be overseen by a safety monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 60-85 years of age at the screening visit and who received AREXVY before.
2. Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccination, laboratory tests, and other study procedures.
3. Individuals willing and able to give an informed consent, prior to screening.
4. Healthy participants as determined by medical history, physical examination, and clinical judgment of the investigator; participants with pre-existing stable medical conditions can be included (a stable medical condition is defined as a disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment).

Please refer to Protocol for full list of Inclusion and Exclusion criteria.

Exclusion Criteria:

1. Acute disease or fever (≥38°C) at time of vaccination. Participants with a minor illness (mild diarrhea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator. For participants with minor illness and/or fever at the time of vaccination, Visit 1 may be rescheduled within the allowed time-window.
2. Recurrent or un-controlled neurological disorders or seizures.
3. Serious or unstable chronic illnesses
4. Any history of dementia or any medical condition that moderately or severely impairs cognition
5. History of a severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccines.

Please refer to Protocol for full list of Inclusion and Exclusion criteria.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and reactogenicity of revaccination with SCB-1019T vaccine | Within 7 days after vaccination
  Proportion of participants with local and systemic solicited AEs
To evaluate the safety and reactogenicity of revaccination with SCB-1019T vaccine | Within 28 days after vaccination
  Proportion of participants with unsolicited AEs
To evaluate the safety and reactogenicity of revaccination with SCB-1019T vaccine | Throughout the study period, from enrollment to 6 months follow up
  Proportion of participants with SAEs, AESIs, MAAEs, AEs leading to early termination from the study

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - AMR Phoenix, Phoenix, Arizona
  - AMR Fort Myers, Fort Myers, Florida
  - AMR Lexington, Lexington, Kentucky
  - AMR Kansas City, Kansas City, Missouri
  - Knoxville, Knoxville, Tennessee